CLINICAL TRIAL: NCT04197388
Title: Inspiratory Muscle Training in Pulmonary Arterial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/CARD/31
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Inspiratory muscle training device — Inspiratory muscle training, 6 cycles of 30 breaths for 12 weeks.

SUMMARY:
Pulmonary arterial hypertension is a rare condition characterised by high blood pressure in the lungs and results in breathlessness and reduced exercise capacity for patients. Previous research has shown weakness in respiratory muscles in these patients that may contribute towards their symptoms. Despite advances in medical therapy, the condition still results in a significant symptom burden.

Inspiratory muscle training is a non-invasive intervention involving a device that provides resistance to the muscles of inspiration and increases their strength.

This study will investigate the benefit of inspiratory muscle training in patients with pulmonary arterial hypertension who are stable on medical therapy for three months. This will be performed as an outpatient and they will then be reviewed following this with assessment of exercise capacity, breathing capacity (spirometry), quality of life, and assessment of neural respiratory drive (the signals from the brain to the muscles controlling breathing).

The study will be based at the Golden Jubilee National Hospital and patients will be recruited from outpatients who are already under the care of the Scottish Pulmonary Vascular Unit.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by pulmonary hypertension specialist with precapillary pulmonary hypertension
* able to give consent
* stable on medical therapy for at least 3 months

Exclusion Criteria:

* significant contribution to pulmonary hypertension from lung disease
* pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Six minute walking distance | 3 months

SECONDARY OUTCOMES:
Quality of life: emPHasis 10 score | 3 months
  emPHasis 10 score
Peak VO2 | 3 months
  Assessed by cardiopulmonary exercise test
VE/VCO2 slope | 3 months
  Assessed by cardiopulmonary exercise test

CONTACTS AND LOCATIONS:
Locations (1):
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No